CLINICAL TRIAL: NCT05586464
Title: The Clinical Trial on the Eradication of Helicobacter Pylori With Bismuth Agent Quadruple and Modified Ban Xia Xie Xin Decoction
Brief Title: Eradication of Helicobacter Pylori With Bismuth Agent Quadruple and Traditional Chinese Medicine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2022-10-05; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-09

CONDITIONS: Helicobacter Pylori Infection; Traditional Chinese Medicine; Eradication
Keywords: Helicobacter Pylori Infection; Traditional Chinese Medicine; Furazolidone; Amoxicillin; Esomeprazole; Pectin bismuth gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese Medicine group (Experimental): Patients in the case group will take Ban xia xie xin Decoction and bismuth quadruplicate for 14 days. H. pylori was rechecked one month after drug withdrawal, and H. pylori clearance rate and adverse reactions were observed in the reorganized patients.
  Ban xia xie xin Decoction includes 10g of banxia, 10g of huangqin, 6g of coptis chinensis, 6g of dried ginger, 6g of ginseng, 6g of roasted licorice, 6g of Chinese jujube. One dose in the morning and one dose in the evening, and take after meals.
  Bismuth quadruplicate includes esomeprazole (nexium, Tablets 20mg/tablet, 20mg bid), amoxicillin ( Tablets 25mg/tablet,100mg bid), furazolidone (Tablets100mg/tablet,100mg bid) and pectin bismuth gel (Gel 150mg/bag, 150mg qid).
  Interventions: Drug: Ban xia xie xin Decoction and bismuth quadruplicate group
- Bismuth quadruplicate group (Active Comparator): Patients in the control group will take bismuth quadruplicate for 14 days. H. pylori was rechecked one month after drug withdrawal, and H. pylori clearance rate and adverse reactions were observed in the reorganized patients.
  Bismuth quadruplicate includes esomeprazole (nexium, Tablets 20mg/tablet, 20mg bid), amoxicillin ( Tablets 25mg/tablet,100mg bid), furazolidone (Tablets100mg/tablet,100mg bid) and pectin bismuth gel (Gel 150mg/bag, 150mg qid).
  Interventions: Drug: Bismuth quadruplicate group

INTERVENTIONS:
Drug: Ban xia xie xin Decoction and bismuth quadruplicate group — Ban xia xie xin Decoction:10g of banxia, 10g of huangqin, 6g of coptis chinensis, 6g of dried ginger, 6g of ginseng, 6g of roasted licorice, 6g of Chinese jujube Bismuth quadruplicate: Esomeprazole (nexium, Tablets 20mg/tablet, 20mg bid), amoxicillin ( Tablets 25mg/tablet,100mg bid), furazolidone (Tablets100mg/tablet,100mg bid) and pectin bismuth gel (Gel 150mg/bag, 150mg qid).
  Other Names: Ban xia xie xin Decoction; Bismuth quadruplicate
  Arms: Traditional Chinese Medicine group
Drug: Bismuth quadruplicate group — Bismuth quadruplicate: Esomeprazole (nexium, Tablets 20mg/tablet, 20mg bid), amoxicillin ( Tablets 25mg/tablet,100mg bid), furazolidone (Tablets100mg/tablet,100mg bid) and pectin bismuth gel (Gel 150mg/bag, 150mg qid).
  Other Names: Bismuth quadruplicate
  Arms: Bismuth quadruplicate group

SUMMARY:
This study is a prospective randomized case-control study. Six hundred patients who were firstly diagnosed as Helicobacter pylori infection will be selected, and then randomly assigned into case group and control group. Patients in control group take bismuth quadruplicate for 14 days. Patients in case group take Ban xia xie xin Decoction and bismuth agent quadruple for 14 days. Exhalation test or stool Helicobacter pylori antigen detection were used to assess the eradication rate of Helicobacter pylori 30 days (the 45th day) after treatment; Adverse reactions were evaluated on the first day (15th day) and the 30th day (45th day) after treatment. The eradication rate of Helicobacter pylori and the adverse drug reactions during the medication will be evaluated. The effect of Ban xia xie xin Decoction and bismuth quadruple based on furazolidone on the eradication of helicobacter pylori infection will be explored.

DETAILED DESCRIPTION:
Helicobacter pylori is a primary carcinogen of gastric cancer. Helicobacter pylori infection rate is about 50% in China. Helicobacter pylori infection should be eradicated unless there are countervailing factors. The bismuth agent quadruple (PPI+bismuth pectin+2 kinds of antibiotics) has eradicated the first line therapy of H. Pylori infection. The rise of antibiotic resistance rate leads to the decline of eradication rate of H. pylori. Traditional Chinese medicine played an important role in the treatment of H. pylori infection. This study explored the application of Ban xia xie xin Decoction and bismuth agent quadruple based on furazolidone in the role of the eradication of H. Pylori infection. This study is a prospective randomized case-control study. Six hundred patients who were firstly diagnosed as Helicobacter pylori infection will be selected, and then randomly assigned into case group and control group. The case group was named as Traditional Chinese Medicine group. Patients in the case group will take Ban xia xie xin Decoction and bismuth quadruplicate for 14 days. The control group was named as bismuth quadruplicate group. Patients in the control group will take bismuth quadruplicate for 14 days. Bismuth quadruplicate includes esomeprazole (nexium 20mg bid), amoxicillin (amoxicillin 1.0 bid), furazolidone (100mg bid) and pectin bismuth gel (150mg qid). Ban xia xie xin Decoction includes 10g of banxia, 10g of huangqin, 6g of coptis chinensis, 6g of dried ginger, 6g of ginseng, 6g of roasted licorice, 6g of Chinese jujube. One dose in the morning and one dose in the evening, and take after meals. Exhalation test or stool Helicobacter pylori antigen detection were used to assess the eradication rate of Helicobacter pylori 30 days (the 45th day) after treatment; Adverse reactions were evaluated on the first day (15th day) and the 30th day (45th day) after treatment. The eradication rate of Helicobacter pylori and the adverse drug reactions during the medication will be evaluated. The effect of Ban xia xie xin Decoction and bismuth quadruple on the eradication of helicobacter pylori infection will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. H. Pylori infection: Carbon13/Carbon14-urea breath test positive or rapid urease test positive or gastric mucosal tissue pathological section positive immunohistochemistry staining or gastric mucosal tissue positive H. pylori culture or fecal Positive detection of H. pylori antigen.
2. No history of H. Pylori infection eradication therapy;
3. Age 18-70 years
4. H.Pylori infection check was completed within 1 month before the start of the study.

Exclusion Criteria:

1. Pregnant or lactating women;
2. There are other serious diseases that affect the evaluation of this study, such as severe coronary heart disease, liver disease, kidney disease, chronic obstructive pulmonary disease, malignant tumor, and psychosocial diseases;
3. History of major or complex gastrointestinal surgery;
4. Those who are allergic to the drugs used in this study;
5. Patients participate other drug studies within 3 months;
6. Patients can not cooperate with the experimenter.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The helicobacter pylori clearance rate in case group and control group. | 45days
  The participants in the case group and the control group were tested for H. pylori after one month of drug withdrawal. If H. pylori was negative, the clearance was successful. The clearance rate of H. pylori was calculated (number of HP negative patients/number of patients included in this group).

SECONDARY OUTCOMES:
Side effects of bismuth quadruple | 45days
  The participants observe whether there are drug-related adverse reactions during and within 30 days after taking the bismuth quadruple. The main side effects of bismuth quadruplex include diarrhea, constipation, abdominal pain, dizziness, headache, rash, insomnia, arthralgia, taste change (oral odor), and others.